CLINICAL TRIAL: NCT04605302
Title: A Prospective Single Blinded, Pilot Study, Comparing a Magnetically Controlled Capsule With or Without a Tether (MCC or MCC-T) With Conventional Upper Endoscopy for the Diagnosis of Patients With Upper Abdominal Symptoms
Brief Title: Comparative Study of MCCE With/Without Tether vs Conventional Upper Endoscopy in Patients With Upper Abdominal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AnX Robotica Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMASS-01
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Upper Gastrointestinal Symptoms

STUDY DESIGN:
Intervention Model Description: Tandem study
Masking Description: Patient blinded to MCC results. EGD assessor blinded to MCC results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm Tandem Study (Experimental): Patients are assigned to swallow a magnetically controlled capsule first then undergo standard gastroscopy
  Interventions: Device: MCC/MCC-T; Device: Standard gastroscopy

INTERVENTIONS:
Device: MCC/MCC-T — Magnetically controlled capsule endoscopy (MCC), with or without tether, is used to visualize the upper gastrointestinal tract
  Other Names: Magnetic controlled capsule endoscopy with/without tether
Device: Standard gastroscopy — Diagnostic endoscopic procedure that visualizes the upper part of the gastrointestinal tract down to the duodenum
  Other Names: EGD

SUMMARY:
A prospective single blinded, tandem study, comparing a magnetically controlled capsule with or without a tether (MCC or MCC-T) with conventional upper endoscopy for the diagnosis of patients with upper abdominal symptoms.

DETAILED DESCRIPTION:
In the US patients commonly undergo esophagogastroduodenoscopy (EGD) for upper abdominal symptoms to try to resolve whether they have gastroesophageal reflux disease or functional dyspepsia, if they are older than the age of 60 with symptoms, or have alarm symptoms such as unexplained weight loss, persistent nausea and vomiting or if they have symptoms that are refractory to acid suppression therapy. Given the increasing burden of digestive disease in the US, the use of EGD is increasing in volume nationwide. EGD usually requires either conscious sedation or monitored anesthesia sedation, which has put an additional cost burden on the healthcare system. Since MCC or MCC-T does not require sedation, it offers an attractive option for both patients and clinicians alike.

The aim of this study is to compare in the same patient the accuracy of the MCC and MCC-T and EGD in patients presenting with upper abdominal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide informed consent
2. Patient has appropriate indications for EGD including symptoms of, but not limited to upper abdominal pain, acid reflux, heartburn, iron deficiency anemia, weight loss, bloating, belching, nausea, vomiting and atypical chest pain.

Exclusion Criteria:

1. Patient with dysphagia.
2. Patient with previous intestinal surgery.
3. Patient with Crohn's disease or other potential obstructive conditions, unless there is a recent CTE, MRE or patency capsule performed to exclude an obstructive lesion that may retain the capsule.
4. Female patient who is pregnant.
5. Patient with implanted medical device that would be potentially affected by magnets or radiofrequency emissions (e.g., pacemakers, implanted cardiac defibrillators).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Number of lesions | 2 days
  Number of lesions found by MCC/MCC-T versus EGD
Number of adverse events | 2 days
  Occurrence and severity of adverse event related to MCC/MCC-T procedure versus EGD procedure

SECONDARY OUTCOMES:
Patient satisfaction score | 2 days
  Patient acceptance of MCC/MCC-T versus EGD (scale of 1 to 10 when 1 is the lowest and 10 is the highest score)

CONTACTS AND LOCATIONS:
Overall Officials: David R Cave, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No